CLINICAL TRIAL: NCT04015999
Title: Microbiota-directed Complementary Food (MDCF) Trial
Brief Title: Community-based Clinical Trial With Microbiota-directed Complementary Foods (MDCFs) Made of Locally Available Food Ingredients for the Management of Children With Primary Moderate Acute Malnutrition
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PR-18073
Record Dates: First submitted 2019-06-23; First posted 2019-07-11 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-06

CONDITIONS: Microbiota; Complementary Food; Nutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention arm (Experimental): MDCF2 with four complementary food ingredients (rationale: lead with evidence from Pre-POC clinical trials to optimize lead microbiota-directed complementary food prototypes for their ability to repair microbiota immaturity and positive effects on growth)
  Interventions: Dietary Supplement: Microbiota Directed Complementary Food (MDCF)
- Control arm (Active Comparator): Rice-lentil based RUSF (rationale: reference standard of care for MAM; based on knowledge of its effects on the gut microbiota or microbiota immaturity)
  Interventions: Dietary Supplement: Ready to Use Supplementary Food (RUSF)

INTERVENTIONS:
Dietary Supplement: Microbiota Directed Complementary Food (MDCF) — MDCF2 with four complementary food ingredients (rationale: lead with evidence from Pre-POC clinical trials to optimize lead microbiota-directed complementary food prototypes for their ability to repair microbiota immaturity and positive effects on growth)
  Arms: Intervention arm
Dietary Supplement: Ready to Use Supplementary Food (RUSF) — Rice-lentil based RUSF (rationale: reference standard of care for MAM; based on knowledge of its effects on the gut microbiota or microbiota immaturity)
  Arms: Control arm

SUMMARY:
Background (brief):

Burden: A total of 52 million children under 5 are suffering from acute malnutrition globally, of whom 33 million have moderate acute malnutrition (MAM). In Bangladesh, more than 2 million children suffer from MAM. According to Bangladesh Demographic Health Survey 2014 26%, 25% and 17% of children aged less than two years are stunted, underweight and wasted respectively.

Knowledge gap: It has been already demonstrated that children with SAM have immature gut microbiota that is partially corrected with treatment. Children with MAM have an increased risk of mortality, infections and impaired physical and cognitive development compared to well-nourished children. Although the global caseload of MAM is much greater than that of SAM, the condition has not received the same level of attention or priority. Through our previous and ongoing research we now know about the members of the gut microbiota that can promote growth in children and also about certain food ingredients that promote the proliferation of such beneficial microbiota. However, this knowledge needs to be applied on a sufficiently powered community-based clinical trial.

Relevance: The rationale for this study is to assess whether long-term administration of complementary food made of locally available food ingredients can stimulate the proliferation of growth promoting members of the gut microbiota and have a positive impact on child growth. Such a food (the microbiota directed complementary food; MDCF-2) has been identified through our recently concluded Pre-proof of concept trial done on children with primary MAM. We would now like to do a clinical community-based trial of this potential MDCF-2 in the management of children with primary MAM.

Hypothesis: Complementary foods made of locally available food ingredients that stimulate the proliferation of growth promoting gut microbiota (MDCF-2) will improve clinical outcomes.

Methods: We will conduct a proof of concept (POC) clinical trial in 12-18 months old children with primary MAM (Weight-for-Length Z-score, WLZ between -2 and -3). This study will be conducted at Bauniabadh, Radda MCH-FP (Maternal and Child Health- Family Planning) clinic, Gabtoli of Mirpur area and possibly at the Special Nutrition Unit run by Terre des Hommes in Kurigram. We will produce MDCF-2 at the icddr,b Food Processing Laboratory or nutrition centre established at the site in sufficient quantities for clinical study. This formulation will be matched in energy density and micronutrient content of ready-to-use supplementary foods (RUSFs) used for MAM in Bangladesh and other countries, and will meet all other requirements for a complementary/supplementary food for 12-18 months old children with MAM. We will test MDCF-2 and the current RUSF standard of care for primary MAM to see the effect on growth, proteomics and metabolomics of an intervention for 12 weeks, with a 4-week post-intervention phase.

Hypothesis to be tested:

In a hypothesis testing research proposal, briefly mention the hypothesis to be tested and provide the scientific basis of the hypothesis, critically examining the observations leading to the formulation of the hypothesis.

Complementary foods made of locally available food ingredients that stimulate the proliferation of growth promoting gut microbiota (MDCF) will provide a new way to improve clinical outcomes, for example by improving growth of children with MAM.

Specific Objectives:

To investigate the efficacy of complementary food made of locally available food ingredients that can stimulate the proliferation of growth promoting gut microbiota (Microbiota-Directed Complementary Food; MDCF-2) in (i) promoting repair of microbiota immaturity (ii) promoting proliferation of beneficial bacteria (iii) improving both ponderal and linear growth in children (iv) improving the metabolomic profile with MAM

DETAILED DESCRIPTION:
Background:

Moderate acute malnutrition (MAM), a major global health problem, is defined as wasting (i.e. weight-for-height between < -2 and -3 Z-scores of the WHO Child Growth Standards) and/or mid-upper-arm circumference (MUAC) greater or equal to 115 mm and less than 125 mm. According to the Global Nutrition Report 2017, 8% or 52 million under-five children were acutely malnourished globally in 2016. Stunting affected 23% or 155 million children. Approximately one in 6 children under 5 years in South Asia suffered from MAM in 2013 (i.e. 17%). These children are at increased risk of severe acute malnutrition (SAM), and have a three times higher risk of mortality from common communicable diseases than the well-nourished peers. Bangladesh has one of the highest childhood malnutrition burdens in the world. According to Bangladesh Demographic Health Survey (BDHS) 2014, the prevalence of stunting among under-five children is 36%, among them 12% suffer from severe stunting (Length-for-Age-Z score, LAZ <-3). Around 15% of children are wasted (Weight-for-Length Z score, WLZ <-2); more than 2 million children suffer from MAM, while 3% or 450,000 children suffer from the deadly form of SAM. Malnutrition costs Bangladesh an estimated US $1 billion a year. According to WHO recommendations, infants and children aged 6-59 months with MAM need to consume nutrient-dense foods to meet their extra needs for weight and height gain and functional recovery. Currently there are no evidence-informed recommendations on the composition of supplementary foods used to treat children with MAM. In situations of food shortage, supplementary foods have been used to treat children with moderate acute malnutrition. Interventions to address under nutrition should therefore include a strong component of MAM management. MAM prevention should be taken into consideration in food security and other development strategies as the situation becomes critical in populations where food insecurity is rampant. Food insecurity has become a worldwide concern due to the increasing number of people who remain undernourished amounting to 842 million, approximately 12% of the total world's population. From the National Micro nutrient Status Survey in Bangladesh which we conducted in 2011-12, severe insecurity of food was found most commonly in slum settlements (17.2 %), compared to 12.3% at the national level, 12% in rural areas and 12.4% in urban areas of the country. Since food insecurity cannot be overcome quite readily, it is important therefore to develop interventions that depend upon locally available food ingredients and are able to harness the beneficial power of the gut microbiota on infant and child growth.

One of the major factors limiting the impact of nutrition intervention is the inability of the malnourished children to increase their intake to meet increased metabolic demands. In collaborative studies between icddr,b and the Gordon Lab at Washington University in St. Louis during the Jump start Phase of the Breast Milk, Microbiota and Immunity (BMMI) Project, we applied Random Forests, a machine-learning-based approach, to bacterial 16S rRNA (ribosomal ribonucleic acid) datasets generated from monthly fecal samples obtained from a birth-cohort of children living in an urban slum of Dhaka, Bangladesh. These children exhibited consistently healthy growth (WLZ -0.32+0.98). Bacterial strains were identified whose proportional representation defines a healthy gut microbiota as it assembles during the first 2-3 postnatal years. In a randomized clinical trial at icddr,b of two therapeutic foods (imported ready-to-use therapeutic food [RUTF (Ready to Use Therapeutic Food), Plumpy'Nut] versus locally prepared rice/lentil-based Khichuri and Halwa) in Bangladeshi children with severe acute malnutrition (SAM), it was observed that the microbiota immaturity is incompletely and only transiently improved, with children remaining markedly stunted and underweight throughout the follow-up period. Bangladeshi children with MAM also exhibited significant microbiota immaturity, although less severe than children with SAM. Microbiota immaturity thus serves as a potential biomarker to identify infants at risk for undernutrition and to monitor treatment and prevention strategies.

Investigators recently developed ready-to-use therapeutic foods using locally available food ingredients-rice, lentil, and chickpeas that are culturally relevant and acceptable. They found through a double-blind RCT (Randomized Controlled Trial) that chickpea-based and rice-lentil-based RUTF were as effective as the commercial peanut based-RUTF and well accepted by children with SAM. Through a combination of the above mentioned RCT and clinical translational studies, they have identified growth promoting age-discriminatory beneficial microbiota and locally available food ingredients that support proliferation of these beneficial microbiota. Besides, results of earlier studies done on gnotobiotic animals in Washington University Centre for Genome Science has led us to suggest that a combination of food ingredients (chickpea, soy flour, peanut and green banana) will be worth studying with respect to the diet's impact on stimulating proliferation of growth-discriminatory microbiota as well as cost and sustainability. To assess the degree to which the results obtained from the gnotobiotic mouse and piglet models translate to humans, investigators recently performed a RRC (Research Review Committee) and ERC (Ethecial Review Committee)approved study, icddr,b protocol (PR-16099) 'Pre-Proof of Concept clinical trials to optimize lead microbiota-directed complementary food (MDCF) prototypes for their ability to repair microbiota immaturity and establish their organoleptic acceptability 'and successfully completed the study. This study was designed to test the effects of three locally produced MDCF prototypes (MDCF-1, MDCF-2 and MDCF-3) and a locally produced rice-lentil-based RUSF. The objective of this pilot study was to demonstrate a Pre-proof of Concept that certain complementary foods would have a beneficial effect on young children suffering from moderate acute malnutrition by stimulating the proliferation of particular members of the gut microbiota that are known for their growth promoting effect. In that pilot study they investigated microbiota-for-age Z score as well as the impact of the proliferation of good members of the gut microbiota on certain body systems. The results of the Pre-POC pilot trial conclusively showed that one of the three microbiota directed complementary foods namely (MDCF-2; composed of a combination of chickpea, soy flour, peanut, green banana, oil, sugar and micronutrients) was associated with increased levels of certain amino acids, that have a key role in development of the long bones, development of the brain and increased production of IGF-1. This was done using the state-of-the-art DNA aptamer based SomaLogic scan. And the results suggest that this candidate MDCF-2 is effective in stimulating the growth of growth promoting members of the gut microbiota, for example Faecalibacterium prausnitzii. Thus, MDCF-2 promotes gut microbiota that induces the hormone insulin-like growth factor 1 (IGF-1), which promotes bone growth and remodelling.

Based on this evidence investigators would now like to do a much larger clinical trial using the most promising MDCF which is MDCF-2 with the primary end point being linear growth. This trial would be on children with primary MAM.

Research Design and Methods Investigators will conduct a clinical trial among 12-18 months old children with primary MAM (WLZ <-2 to -3).

Study design: Randomized controlled intervention trial. Study site: This study will be conducted at Bauniabadh, RADDA MCH-FP (Maternal and Child Health - Family Planning) clinic in Mirpur area and Gabtoli of Dhaka city, and possibly at the Special Nutrition Unit run by Terre des Hommes in Kurigram.

Study participants: The study participants will be 12-18 months old children of either sex with MAM (WLZ <-2 to -3).

Initial screening and enrolment: Children will be screened and enrolled through household surveys by Field Research Assistants (FRAs) following pre-specified inclusion criteria. Fulfilling the enrollment criteria and upon receiving the consent for study participation from the parents or legal guardians, the children with the respective mother/caregiver will be enrolled and randomly assigned to one of the two arms according to computer-generated random numbers. The code of assigned type of diet will be kept in closed opaque envelopes for each individual, and will be opened only when the caregiver signs the consent form.

Study design:

Arm 1 - Rice-lentil based RUSF (rationale: reference standard of care for MAM; based on knowledge of its effects on the gut microbiota or microbiota immaturity) Arm 2 - MDCF2 (Microbiota Directed Complementary Food 2) with four complementary food ingredients (rationale: lead with evidence from Pre-POC clinical trials to optimize lead microbiota-directed complementary food prototypes for their ability to repair microbiota immaturity and positive effects on growth) Fecal sample collection Weekly fecal samples (1-2g) will be collected within 30 minutes of excretion (at home and transported back to the icddr,b) using the liquid nitrogen containing dry shipper. Specimens will be stored at -80°C before being sent to the Gordon Lab analysis of microbiota maturity (measured before, during and after cessation of treatment with MDCF and RUSF) and PCR (Polymerase Chain Reaction)-based assessment of enteropathogen burden in fecal samples (measured before and after MDCF treatment).

1-2 gm of fecal samples will be collected from each child at enrollment, weekly during the 1st month of intervention, and 4 weekly during the 2nd and 3rd month of intervention and at the end of post-intervention phase. Assuming 62 study participants /arm, a total of 992 fecal specimens will be collected in this study. 2 gm of faecal samples will be collected from mothers at the time of enrollment.

Urine sample collection 2 mL of urine samples will be collected from each child at enrollment, one week after enrollment and monthly once in the intervention and post-intervention phases. Assuming 62 study participants /arm, a total of 744 urine samples will be collected in this study. 5 mL of urine samples will be collected from mothers at the time of enrollment.

Blood sample collection 2 mL of blood samples each will be collected from each child prior to intervention, end of first month of intervention and just after the intervention is complete. A total of 372 plasma samples will be collected in this study. 5 mL of blood samples will be collected from mothers at the time of enrollment.

Maternal nutritional status is associated with child nutritional status, as shown through the results of our eight country MAL-ED (Malnutrition and Enteric Diseases) study. In addition, neonatal and other maternal factors were early determinants of lower length-for-age, and their contribution remained important throughout the first 24 months of life.9 The other maternal factors, investigators believe, would include maternal gut microbiota as well as maternal blood amino acid profile. Initiatives to address childhood stunting should also consider improvements to the composition of complementary foods (i.e., higher protein) and strategies to reduce gut pathogen exposure. As such, they will record maternal height and weight. In order to understand the biological state of nutrition of the mother, enrolment samples of stool, blood and urine will be asked of the mother. These samples will be analyzed for gut microbiota, and proteomics, and the results correlated with those of the enrolled children.

Feeding sessions The children and mothers/caregivers will be requested to come to the nutrition centers established at the sites preferably between 9-11 am and 3-5 pm on day 1. The mothers will be requested not to give any food and breast milk in the 2 hours preceding the observed meal time. The child will be offered 25 grams of MDCF or RUSF as decided by random allocation in each of the two meals between 9-11 am and 3-5 pm. The mothers will be asked to spoon feed the pre-weighed diets to their children until s/he refuses to eat, as described below. After a two-minute pause, the same diet will be offered a second time until s/he refuses again. After a second two-minute pause, the diet will be offered a third time until refused again. After this third refusal, the feeding episode will be considered as 'terminated'. The duration of the feeding (excluding the intervening 'rest periods') will be recorded by stopwatch, and the total duration of the feeding will be noted. This feeding episode will last for maximum 60 minutes. Measured volumes of plain water will also be given and the amount of water taken during this meal period of 60 minutes will be measured. The feeding episode will take place under the direct supervision of trained study personnel. Children will be considered as refusing further intake if they move their head away from the food, cry, clamp the mouth or clinch the teeth, or become agitated, spit out the food or refuse to swallow. The amount of MDCF/RUSF actually ingested will be calculated by subtracting the left over from the offered amount. Pre-weighed napkins will be provided; any food that is regurgitated, vomited or spilled will be swabbed, weighed and subtracted from the amount offered. The amount of consumed food (g), energy (kcal) and category of acceptability will be analyzed. The enrolled children will be monitored daily by Field Research Assistants for any possible side effects/adverse events (e.g. rash, urticaria due to food allergy or any significant changes in clinical status) for a week. If any side effects/adverse events are observed, they will be treated according to standard of care. A standardized production procedure will be followed to control the quality of RUSF and MDCF following international standard protocol. RUSF and MDCF will be prepared at the food processing laboratory. Preparation of food under different steps, that is, roasting, particle size reduction, homogeneous blending, and supplying to the nutrition centres will be monitored by icddr,b investigators. Food will be prepared everyday to ensure that no unexpected contamination and nutrient losses occur during preparation. Although raw food ingredients will be very carefully procured from the local market and stored in reasonable quantities, investigators will prepare, dispense, and feed the children the same day the MDCF and RUSF are prepared. Every child will be offered 25gm of the diet twice daily at the feeding center for the first 4 weeks. In the following month, the child will be offered 25gm of the diet at the feeding center and additional 25gm will be provided in a clean container to feed at home. In the third month, two separate containers containing 25gm diet will be provided every day to each enrolled child at participant's home.

In this study nutritional status will be assessed through anthropometry, comparing with WHO growth reference standards. At the beginning of the study, information will be sought on the demographic characteristics (families' wealth, standard of housing, family structure and parental characteristics etc.), and FRAs will record the children's weight using a digital scale with 2g precision (Seca, model 728, Germany), length (using infantometer, Seca, model 416, Germany), and mid upper-arm circumference to the nearest mm (using a non-stretch insertion tape). Anthropometrics will be done according to the standard procedures and all measurements will be taken thrice and the middle one will be recorded.

All interventions in each study will be administered to children at the Mirpur health clinic/RADDA clinic or in Kurigram. Mothers/primary caregivers will be advised to maintain their child's current dietary and breastfeeding practices.

Investigators will complete enrollment within 12 months and the follow up as well as data analysis within an additional 6 months. However, this trial on primary MAM will continue simultaneously with the other clinical trial on Post SAM-MAM that will have a longer period of duration.

Recruitment, Screening and Consenting Census, screening, enrolment of study participants will be done in the catchment areas of the sites in Dhaka city and in Kurigram. Parents of children who meet the MAM criteria (for Primary MAM trial) will be approached about enrollment into the study. A Field Research Assistant will explain the study in detail, answer any questions from the parent(s), and invite the parent(s) to enroll the child in the study.

At the beginning of the study, information will be sought on the demographic characteristics (families' wealth, standard of housing, family structure and parental characteristics etc.), and FRAs will record the children's weight using a digital scale with 2 g precision, length (using infantometer,), and mid-upper-arm circumference to the nearest mm. Study participants will be asked to come directly to the nutrition center for nutritional therapy.

Preparation of MDCF 2 and RUSF Based on compatible combinations of complementary food ingredients identified in the Pre-POC study described above, MDCF2 as well as Rice-lentil RUSF will be produced at the icddr,b Food Processing facility in Mirpur and in Kurigram (to be established in both places) in sufficient quantities for clinical study. The two diets will be matched in energy density and micronutrient content. The energy density of MDCF is 125 kcal/25 g (per serving), and caloric distribution is targeted to be 45-50 percent from fat and 8-10 percent from protein. Experiments in development of the MDCF prototypes and assessment of the organoleptic properties have been done during the Pre-POC clinical trial. After receiving the raw materials (rice/lentil/chickpea) the foreign materials/grains or seeds (if there is any) will be taken out, and then in an open pan the raw materials will be roasted. The temperature will be maintained at 120-130°C for roasting. Usually it takes 8-10 minutes for roasting 100g of each raw material. Continuous stirring is essential to ensure roasting of single seeds/grains. After completion of roasting it will be kept aside for cooling and then will be grinned. Finally the pre-weighed premix powder will be added. The processing of whole green banana for inclusion in MDCF2 is different from the other ingredients. Green banana with skin will be placed in a deep pan in boiling water (100°C-110°C) and boiled for about 17-20 minutes until they are cooked and tender. The skin of the green banana will be peeled off and the edible white part would be taken and grated into small pieces. Then they will be taken in a pot and allowed to cool. The small pieces of banana will be smashed with spoon/hand crusher. The weights of all other ingredients will be recorded. Recipes will be produced in small batches by mixing all ingredients in an electric blender. A small amount (1 percent) of soy lecithin shall be added to the recipe in order to improve the consistency and prevent oil separation.

Anthropometry The age of the child will be verified against documentation (birth certificate or immunization card, if available) or caregiver's report of the child's birth date. Length will be measured by a infantometer sensitive to 0.1 cm. Body weight will be measured by a balance sensitive to 2g. Length-for-age (LAZ), weight-for-length (WLZ) and Weight-for-Age (WAZ) Z-scores will be calculated following the Multicentre Growth Reference Study (MGRS) WHO (World Health Organization) growth standards. Edema will be examined by pressing the upper side of both feet for 3 seconds. Mid-upper arm circumference (MUAC) will be measured using MUAC tape (UK). Regular standardization of the measuring equipments will be done using standards.

Analyses of plasma and fecal samples Plasma samples collected from this trial will be sent to Dr Jeffrey Gordon's lab in the Center for Genome Sciences and Systems Biology at Washington University in St. Louis. Advanced mass spectroscopic- and immunoassay-based methods will be used to obtain new knowledge about the role of gut microbiota immaturity and the effects of attempting acute repair of this immaturity with lead microbiota-directed complementary food (MDCF) on biomarkers and mediators of healthy growth. Comparisons will be made with the control group (i.e., those consuming reference RUSF standard). Targeted Ultra Performance Liquid Chromatography-Mass Spectrometry (UPLC-MS) and Gas Chromatography-Mass Spectrometry (GC-MS) will be used to profile analytes of specific interest in plasma and/or fecal samples including bile acids and short chain fatty acids (SCFAs); markers of mitochondrial function (e.g., β-hydroxybutyrate, acylcarnitines/acylCoAs, TCA cycle intermediates); amino acids in serum plus fecal samples [branch chain amino acids, tryptophan and tryptophan metabolites related to growth and inflammatory status, including those produced by bacterial tryptophan metabolism (e.g. indole acetic acid derivatives)]. Key mediators/biomarkers of linear growth (e.g., growth hormone and IGF-1), energy utilization (insulin, leptin), and bone biology [IL-6 (Interleukin-6), osteoprotegerin, the C-terminal peptide of type I collagen (CTX, a marker of osteoclast activity/bone resorption), and the amino-terminal propeptide of Type 1 procollagen (P1NP, a marker of osteoblast activity/bone formation)], and systemic inflammation (CRP, AGP) will be quantified using established ELISA/Luminex assays. Proteins in blood will be identified using the SOMAlogic scan that permits identification of more than 1300 different proteins. The proteomic study done on plasma samples from children with SAM in our previous Pre-POC trial done in Dhaka has already demonstrated a number of significant and clinically relevant associations between certain proteins and clinical phenotypes using the SOMAlogic scan.

Information gathered will be used to select human fecal samples for transplantation into germ-free animals in the Gordon Lab in St Louis; these animals, who will be fed the diets of their human microbiota donors, will be used to further characterize the mechanisms that link MDCF prototypes, the gut microbiota, and host physiology/metabolism. In addition, these plasma and fecal biomarkers will be used to determine that MDCF promotes repair of microbiota immaturity and improves biological state in children.

Sample Size Calculation In the pre-POC trial of different MDCFs, the baseline weight-for-length Z score of children who received MDCF2 was -2.2 and after one month of supplementation was -1.7. If it is considered the WLZ -2 at baseline and -1.7 at end line, pooled SD (Standard Deviation)as 0.53 then the sample size is 49 in each arm at 80% power and 5% level of significance.

With 20% attrition 62 children will be required to be enrolled in each arm. Therefore, for the Primary MAM trial, 62 children will receive MDCF2 and 62 children will receive Rice-lentil RUSF.

Data Analysis The two groups of children with MAM will be compared at baseline and at different time points. All analytes mentioned in the section Analyses of plasma and fecal samples' will be compared between MDCF2 and RUSF groups.

Data Safety Monitoring Plan (DSMP) Data collection tools for this study will include case report forms, laboratory worksheets and source documentation. Complete source documentation (study visits, laboratory reports, etc.) will be kept for each study participant in individual study charts. All laboratory specimens, reports, study data collection and administrative forms will be identified by coded number to maintain study participant confidentiality and to enable tracking throughout the study.

Forms, lists, logbooks, appointment books, and any other listings that link study participant ID (Identification) numbers to other identifying information will be stored in a separate, locked file in an area with limited access. All information regarding study participants will be kept in password-protected computer files or in locked file cabinets that can be accessed only by authorized study personnel. Chart information and information from study records will not be released without written permission from the study participant's parent(s). However, records may be reviewed by representatives from the Research Review Committee and Ethical Review Committee of icddr,b.

The study investigators are responsible for ensuring complete and accurate documentation for the study and for each study participant, including: medical records, records detailing each study participant's progress through the study, laboratory reports, Case Report Forms (CRFs), signed informed consent forms, correspondence with IRB (Institutional Review Board ), adverse event reports, and information regarding participant discontinuation and completion of the study. All required data will be clearly and accurately recorded in the CRFs by authorized study personnel. Only designated study-site personnel who have received appropriate training will record or change data in a CRF. The investigators are responsible for procuring the data and for quality of data recorded in the CRFs. Data entry and management will be performed at icddr,b.

Ethical Assurance for Protection of Human rights The study will be started after obtaining IRB approval by the icddr,b Research Review Committee and Ethical Review Committee. Before enrolment in the study, informed written consent will be taken from the legal guardian of the study participants. The privacy, anonymity and confidentiality of data/information identifying the study participants will be strictly maintained. Personal identifications taken during enrolment and other study procedures will be kept under lock and key. None other than the study personnel will have access to information of personal identification and other sensitive information.

Expected risks/adverse events for this protocol are those related to blood sample collection, fecal sample collection and feeding of microbiota directed complementary food. None of these qualify as a serious adverse event (SAE). Expected Adverse Events (EAEs) related to blood draw are as follows:

* discomfort
* pain
* introduction of infection
* bleeding
* fainting or bruising

  * Precaution will be taken to avoid introduction of infection by disinfecting the site of venipuncture and using sterile equipment
  * The risk of bleeding and bruising will be minimized by immediate application of pressure after venipuncture
  * The participant (child) will be in the sitting or supine position during blood draws to avoid injuries from fainting

All possible adverse events will be treated appropriately. These will include:

* Vomiting
* Diarrhoea
* Skin rash
* Urticaria from food allergy
* Abdominal distension
* Pain abdomen Assessment of Adverse Events Both serious and non-serious adverse events will be assessed for severity; relationship to study participation; actions taken; and outcomes. All SAEs will be reported to the ERC of icddr,b within 24 hours of the site's awareness of the event that will in turn be distributed to the sponsor. This will be done by direct telephone communication, fax or e-mail.

Each category for AE assessment will be coded according to the following grading systems:

Severity:

1. Mild
2. Moderate
3. Severe

Relationship to Study Participation:

1. Definitely related: Clear cut temporal association, no other possible cause
2. Possibly related: Less clear cut temporal association, other causes possible
3. Unrelated: Independent of study, evidence exists that event is definitely related to another etiology

Actions:

None Remedial therapy (more than one dose of medicine required) Permanently discontinued from study participation Hospitalization Other Use of Animals Not applicable Collaborative Arrangements This project is a collaborative effort between the investigators in the Washington University School of Medicine and the International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b). The clinical work, field activities will be undertaken in Dhaka, Bangladesh, under the direct supervision of the Principal Investigator whereas the laboratory analyses will be conducted at the Gordon Lab at Washington University in St. Louis. All research units and the collaborating investigators have long histories of international collaborations. All investigators have communicated during development of this project and are committed to its successful implementation.

Facilities Available icddr,b has a well equipped Food Processing Lab that will facilitate preparations of diet recipes. A number of project offices are located in Mirpur. More importantly, an excellent rapport has been established with the community. The community elite and elders are invited every year to a dissemination meeting so that they are aware of the research being conducted.

Center for Genome Sciences, Washington University in St. Louis:

ELIGIBILITY:
Inclusion Criteria:

* Parent(s) willing to sign consent form
* Child age 12-18 months and no longer exclusively breast fed
* WLZ (<-2 to -3) without bilateral pedal edema at the time of randomization
* Parent(s) willing to bring the child to the feeding center twice daily for 4 weeks for nutritional therapy, once daily for next 4 weeks and provide feeding once daily at home for 4 weeks and twice daily for next 4 weeks.
* The informed consent document will explicitly request permission to use the collected fecal samples for future studies, including but not limited to culturing component bacterial strains

Exclusion Criteria:

* Medical conditions: Children with tuberculosis (diagnosis based on WHO 2014 guidelines which have been incorporated in the national TB control guidelines of Bangladesh). The guidelines depend upon the following five diagnostic principles (three out of five should be positive): 1. Specific symptoms of TB, 2. Specific signs, 3. Chest X-ray, 4. Mantoux test, and 5. History of contact. 10 or any congenital/acquired disorder affecting growth i.e. known case of trisomy-21 or cerebral palsy; children on an exclusion diet for the treatment of persistent diarrhea; having known history of soy, peanut or milk protein allergy
* Antibiotic use within the last 15 days
* Receiving concurrent treatment for another condition
* Severe anemia (<8mg/dl) will be assessed by Hemocue (Model no. Hemocue Hb 301)
* Failure to obtain informed written consent from parents or caretakers

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-06-28 (Estimated); Study Completion 2021-06-28 (Estimated)

PRIMARY OUTCOMES:
Change in Ponderal growth | At the enrollment (day1), every 15 days during the 3 months of intervention phase and at the end of 1 month of follow up phase by anthropometry
  Rate of weight gain of the enrolled participants
Change in Linear growth (LAZ), | At the enrollment (day1), every 15 days during the 3 months of intervention phase and at the end of q month of follow up phase by anthropometry
  Rate of skeletal human growth
Change in Proteomic profile | A total of 3 Plasma samples will be collected, just before the start of intervention phase, at the end of first month of intervention phase and just after the completion of 3rd month.
  Information about all proteins that are made in blood, other body fluids, or tissues, at certain times. It will be assayed by Somalogic scan.
Change in Morbidity | Data will be collected every day during the 3 months of intervention phase and once at the end of 1 month of follow up phase.
  Refers to having a disease or a symptom of disease. It will be assessed by taking morbidity data.
Change in microbiota-for-age Z score | At the enrollment, at the beginning of the intervention phase, weekly during the 1st month of intervention, at the end of 2nd and 3rd months of intervention and at the end of 1 month of follow up phase.
  Bacterial species whose proportional representation define a healthy gut microbiota as it assembles during the first two postnatal years of life.'Microbiota-for-age-Z-score' compares development of a child's fecal microbiota relative to healthy children of similar chronologic age.

CONTACTS AND LOCATIONS:
Overall Officials: Tahmeed Ahmed, PhD, MBBS, Principal Investigator — Senior Director, Nutrition & Clinical Services Division, icddr,b; Munirul Islam, PhD, MBBS, Study Chair — Scientist, Nutrition and Clinical Services Division, icddr,b; Mustafa Mahfuz, MPH, MBBS, Study Chair — Associate scientist, Nutrition and Clinical Services Division, icddr,b; Sayeeda Haque, MPH, MBBS, Study Chair — Associate Scientist, Consultant Physician, Nutrition Ward, Nutrition & Clinical Services Division, icddr,b; Ishita Mostafa, MPH, MBBS, Study Chair — Research Investigator, Nutrition & Clinical Services Division, icddr,b; Imteaz Mahmud, MBBS, Study Chair — Research Fellow, Nutrition & Clinical Services Division, icddr,b; Nurun Nahar Naila, MPH, MBBS, Study Chair — Assistant scientist, Nutrition & Clinical Services Division, icddr,b
Locations (1):
- Icddr,B, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Hawkes C. Global nutrition report 2017: Nourishing the SDGs. Development Initiatives; 2017.
- [Background] James P, Sadler K, Wondafrash M, Argaw A, Luo H, Geleta B, Kedir K, Getnet Y, Belachew T, Bahwere P. Children with Moderate Acute Malnutrition with No Access to Supplementary Feeding Programmes Experience High Rates of Deterioration and No Improvement: Results from a Prospective Cohort Study in Rural Ethiopia. PLoS One. 2016 Apr 21;11(4):e0153530. doi: 10.1371/journal.pone.0153530. eCollection 2016. PMID 27100177
- [Background] 3. National Institute of Population Research and Training (NIPORT), Mitra and Associates, and ICF International. 2016. Bangladesh Demographic and Health Survey 2014. Dhaka, Bangladesh, and Rockville, Maryland, USA: NIPORT, Mitra and Associates, and ICF International.
- [Background] 4. Save the children (2015), malnutrition in Bangladesh: Harnessing social protection for the most vulnerable (2015).
- [Background] Blanton LV, Barratt MJ, Charbonneau MR, Ahmed T, Gordon JI. Childhood undernutrition, the gut microbiota, and microbiota-directed therapeutics. Science. 2016 Jun 24;352(6293):1533. doi: 10.1126/science.aad9359. PMID 27339978
- [Background] Subramanian S, Huq S, Yatsunenko T, Haque R, Mahfuz M, Alam MA, Benezra A, DeStefano J, Meier MF, Muegge BD, Barratt MJ, VanArendonk LG, Zhang Q, Province MA, Petri WA Jr, Ahmed T, Gordon JI. Persistent gut microbiota immaturity in malnourished Bangladeshi children. Nature. 2014 Jun 19;510(7505):417-21. doi: 10.1038/nature13421. Epub 2014 Jun 4. PMID 24896187
- [Background] Choudhury N, Ahmed T, Hossain MI, Islam MM, Sarker SA, Zeilani M, Clemens JD. Ready-to-Use Therapeutic Food Made From Locally Available Food Ingredients Is Well Accepted by Children Having Severe Acute Malnutrition in Bangladesh. Food Nutr Bull. 2018 Mar;39(1):116-126. doi: 10.1177/0379572117743929. Epub 2017 Dec 19. PMID 29258336
- [Background] Yan J, Herzog JW, Tsang K, Brennan CA, Bower MA, Garrett WS, Sartor BR, Aliprantis AO, Charles JF. Gut microbiota induce IGF-1 and promote bone formation and growth. Proc Natl Acad Sci U S A. 2016 Nov 22;113(47):E7554-E7563. doi: 10.1073/pnas.1607235113. Epub 2016 Nov 7. PMID 27821775
- [Background] MAL-ED Network Investigators. Childhood stunting in relation to the pre- and postnatal environment during the first 2 years of life: The MAL-ED longitudinal birth cohort study. PLoS Med. 2017 Oct 25;14(10):e1002408. doi: 10.1371/journal.pmed.1002408. eCollection 2017 Oct. PMID 29069076
- [Background] 10. World Health Organization. World health statistics 2016: monitoring health for the SDGs sustainable development goals. World Health Organization; 2016 Jun 8.
- [Background] de Onis M, Garza C, Victora CG, Onyango AW, Frongillo EA, Martines J. The WHO Multicentre Growth Reference Study: planning, study design, and methodology. Food Nutr Bull. 2004 Mar;25(1 Suppl):S15-26. doi: 10.1177/15648265040251S103. PMID 15069916
- [Derived] Chen RY, Mostafa I, Hibberd MC, Das S, Mahfuz M, Naila NN, Islam MM, Huq S, Alam MA, Zaman MU, Raman AS, Webber D, Zhou C, Sundaresan V, Ahsan K, Meier MF, Barratt MJ, Ahmed T, Gordon JI. A Microbiota-Directed Food Intervention for Undernourished Children. N Engl J Med. 2021 Apr 22;384(16):1517-1528. doi: 10.1056/NEJMoa2023294. Epub 2021 Apr 7. PMID 33826814
- [Derived] Mostafa I, Nahar NN, Islam MM, Huq S, Mustafa M, Barratt M, Gordon JI, Ahmed T. Proof-of-concept study of the efficacy of a microbiota-directed complementary food formulation (MDCF) for treating moderate acute malnutrition. BMC Public Health. 2020 Feb 17;20(1):242. doi: 10.1186/s12889-020-8330-8. PMID 32066412